CLINICAL TRIAL: NCT03225495
Title: Éxito a Corto Plazo de Los Implantes Ultra-estrechos (2,75 mm) en comparación Con Implantes de Plataforma Regular (4,3 mm) Que Requieren regeneración ósea Vestibular simultánea. Ensayo clínico Aleatorizado
Brief Title: Comparison Between Ultra-narrow Diameter Implants (2,75 mm) Without Bone Regeneration Versus Standard Diameter Implants (4,3 mm) in Combination With Bone Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Collaborators: Adin Implants (Unknown); Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Rui Figueiredo, PhD - Assitant Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39/2016
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Dental Implant; Narrow Implant; Implant Fracture; Guided Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Implant (Active Comparator)
  Interventions: Procedure: Standard implant
- Ultra-narrow Implant (Experimental)
  Interventions: Procedure: Ultra-narrow implant

INTERVENTIONS:
Procedure: Standard implant — Arm - Standard Implant: implant placement in combination with guided bone regeneration;
  Arms: Standard Implant
Procedure: Ultra-narrow implant — Arm - Ultra-narrow implant: implant placement without guided bone regeneration
  Arms: Ultra-narrow Implant

SUMMARY:
The main target of the study is to compare ultra-narrow diameter implants (2.75 mm) without bone regeneration versus standard diameter implants (4.3 mm) in combination with bone regeneration. To do so, patients with missing upper central incisors, canines, first or second premolars with alveolar ridges of 6 - 8 mm of thickness will be restored with dental implants. Cone beam computed tomographic examination and clinical values will be registered before and after the surgical procedure at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* One missing teeth in position: upper central incisor, canine or premolar
* alveolar ridge thickness of 6 - 8 mm
* alveolar ridge height of ≥ 10 mm

Exclusion Criteria:

* Missing data
* ASA ≥ III

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Success | 12 months
  According to criteria described by Albrektsson et al. 1986

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Odontològic - Universitat de Barcelona, L'Hospitalet de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: Undecided